CLINICAL TRIAL: NCT02266173
Title: Post-Marketing Surveillance of Perjeta in Breast Cancer
Brief Title: Observational Study of Pertuzumab Safety in Participants With Breast Cancer
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML29299
Record Dates: First submitted 2014-09-30; First posted 2014-10-16 (Estimated); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — pertuzumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Pertuzumab: Participants for whom the treating physician has decided to administer pertuzumab according to standard of care and in line with the current summary of product characteristics (SmPC)/local labeling, will be observed.
  Interventions: Drug: Pertuzumab

INTERVENTIONS:
Drug: Pertuzumab — Study protocol does not specify/enforce any particular dosage regimen. Pertuzumab will be administered according to standard of care and in line with current SmPC/local labelling.
  Other Names: Perjeta

SUMMARY:
This Phase IV, prospective, multicenter, non-interventional study (regulatory post-marketing surveillance) will evaluate the safety of pertuzumab in approximately 1000 participants with metastatic or locally unresectable recurrent breast cancer who have never received chemotherapy or anti-human epidermal growth factor receptor 2 (HER2) therapy for their metastatic disease with HER2 positivity in Korea. Participants who are administered with pertuzumab according to medical opinions of the doctor in charge of surveillance will be registered for this study and treated with pertuzumab under the approval conditions of the product in Korea.

ELIGIBILITY:
Inclusion Criteria:

* Participants with metastatic or locally unresectable recurrent breast cancer who have never received chemotherapy or anti-HER2 therapy for metastatic disease with HER2 positivity
* HER2-positive, locally advanced, inflammatory, or early stage breast cancer (greater than [>]2 centimeters [cm] in diameter) participants who have never received chemotherapy and surgery for breast cancer

Exclusion Criteria:

* Hypersensitivity for pertuzumab (Perjeta) or any of its excipients
* Contraindications to Perjeta according to SmPC
* Pregnancy and lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants with metastatic or locally unresectable recurrent breast cancer and have never received chemotherapy or anti-HER2 therapy for metastatic disease with HER2 positivity.
Sampling Method: Non-Probability Sample
Enrollment: 1130 (Actual)
Dates: Start 2015-02-05 (Actual); Primary Completion 2021-03-08 (Actual); Study Completion 2021-03-08 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | Baseline up to approximately 6 years

SECONDARY OUTCOMES:
Percentage of Participants With Overall Response as Determined Using Response Evaluation Criteria in Solid Tumors (RECIST) | Baseline until disease progression or death, whichever occurs earlier (assessed up to approximately 6 years)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (37):
- South Korea (37):
  - Inje university Haeundae Paik Hospital, Busan
  - Pusan National University Hospital, Busan
  - Kosin University Gospel Hospital, Busan
  - Kyungpook National University Chilgok Hospital, Daegu
  - Keimyung University Dongsan Medical Center, Daegu
  - Chungnam National University Hospital, Daejeon
  - National Health Insurance Service Ilsan Hospital, Gyeonggi-do
  - Hallym University Sacred Heart Hospital, Gyeonggi-do
  - Soonchunhyang University Bucheon Hospital, Gyeonggi-do
  - St. Vincent's Hospital, Gyeonggi-do
  - Ajou University Medical Center, Gyeonggi-do
  - The Catholic University of Korea Bucheon St. Mary's Hospital, Gyeonggi-do
  - Pusan National University Yangsan Hospital, Gyeongsangnam-do
  - Catholic Univ. of Incheon St.Mary's Hospital, Incheon
  - Inha University Hospital, Incheon
  - Gil Hospital. Gachon University, Incheon
  - Catholic Kwandong University International St. Mary'S Hospital., Incheon
  - Chonnam National University Hwasun Hospital, Jeollanam-do
  - Wonkwang University School of Medicine & Hospital, Jeonlabuk-do
  - Seoul National University Bundang Hospital, Seongnam-si
  - Samsung Medical Center, Seoul
  - Inje University, Sanggye-Paik Hospital, Seoul
  - Korea Cancer Center Hospital of Korea Institute of Radiological and Medical Sciences, Seoul
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Konkuk University Medical Center, Seoul
  - Gangdong Kyung Hee University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Gangnam Severance Hospital, Seoul
  - Seoul St Mary's Hospital, Seoul
  - ChungAng University Hospital, Seoul
  - Yeouido St. Mary's Hospital, Seoul
  - Ewha Womans University Mokdong Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - SMG-SNU Boramae Medical Center, Seoul
  - Ulsan University Hosiptal, Ulsan